CLINICAL TRIAL: NCT05522452
Title: Comparison of Synchronous Telerehabilitation and Face to Face Method for Improving Upper Extremity Functions in Children With Hemiparetic Cerebral Palsy
Brief Title: Synchronous Telerehabilitation vs Face to Face Method for Upper Extremity Functions in Children With Hemiparetic CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Polen Altun, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PhD thesis
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): The telerehabilitation group will participate in the treatment in their homes. While the participants are performing the activities in their own homes, applications will be made via webcam-based software (Zoom) and synchronous access via video and audio from the physiotherapist's computer screen. The activities determined by the physiotherapist will be directed to the family, and the activities will be adapted and implemented according to the child's needs and functional level.
  Physiotherapy program will include the following applications:
  * Tone regulation
  * Active stretching and strengthening exercises
  * Gross and fine motor activities to improve bilateral hand use
  * Daily living activities to improve upper extremity functional skills such as dressing, eating, and buttoning.
  * Arts and crafts activities
  Interventions: Other: Telerehabilitation
- Face to face group (Active Comparator): The face-to-face group will be treated in the clinic. To this group; The activities determined by the physiotherapist will be applied face to face.
  Physiotherapy program will include the following applications:
  * Tone regulation
  * Active stretching and strengthening exercises
  * Gross and fine motor activities to improve bilateral hand use
  * Daily living activities to improve upper extremity functional skills such as dressing, eating, and buttoning.
  * Arts and crafts activities
  Interventions: Other: Face to face rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Telerehabilitation program: Intervention will be applied by video interview for 12 weeks, 2 days a week, 45 minutes a day through the Zoom application. The application is free and can be installed on desktop or laptop computers, tablets and smartphones. The content of the activities to be done for that session by phone call to the parent before the interventions; Information will be given about the preparations such as keeping the materials on the table, suitable environment for that week's session and camera angle. Instructions and tips for parent support during the intervention will be given before and during the session. Intervention will be focused on upper extremity skills and activities of daily life of the individuals.
  Arms: Telerehabilitation group
Other: Face to face rehabilitation — Face to face program: Intervention will be applied by physiotherapist for 12 weeks, 2 days a week, 45 minutes a day in clinic. Intervention will be focused on upper extremity skills and activities of daily life of the individuals.
  Arms: Face to face group

SUMMARY:
The aim of this study is to investigate the effectiveness of synchronous telerehabilitation on improving upper extremity function in children with hemiparetic cerebral palsy.

DETAILED DESCRIPTION:
46 children with hemiparetic cerebral palsy who meet the inclusion criteria and agree to participate in the study will be included. The participants will be randomly divided into two groups. The groups are: a) the synchronous telerehabilitation group; b) face to face rehabilitation group. Both groups will receive physiotherapy 2 days a week (1 session of 45 minutes) for 12 weels, for a total of 24 sessions. Evaluations will be made at baseline and the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of confirmed hemiparetic cerebral palsy
* Manual Ability Classification System ≤ 3
* Age between 6 and 18
* Absence of major visual and/or auditory deficits
* Sufficient cooperation to comprehend and complete the test procedure and participate in treatment
* Family members being active mobile phone or computer and internet users

Exclusion Criteria:

* Seizures uncontrolled by therapy
* Surgery and/or botulinum toxin-A injections in the upper limb within 6 months prior to the baseline assessment
* Having a disabling behavioral disorder to treatment
* Family's discontinuation of treatment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Quality of Upper Extremity Skills Test (QUEST) | 12 weeks
  It is used to evaluate the upper extremity motor functions of children. QUEST is a test that evaluates the quality of movement and dexterity of the child with SP. QUEST is concerned with how the child does the activity he or she can do. Examines the quality of upper limb skills in 7 sections. The highest score is 100, the lowest score is 50
The Selective Control of the Upper Extremity Scale (SCUES) | 12 weeks
  This test was developed to evaluate the selective motor control of the upper extremity. It is a very practical and useful video-based assessment tool that can be applied in less than 15 minutes. No special equipment is required other than a video camera. It offers the opportunity to evaluate the selective movements of the shoulder, elbow, forearm, wrist and fingers for both right and left extremities. The person administering the test passively shows the participant the movements they are asked to do. Then the participant is asked to actively perform the movement shown. While performing the participant movements; Head, trunk and other extremity movements are taken with a video camera to provide the opportunity to observe. The degree of selective motor control is determined as 0-3 points for each joint, depending on the person's ability to perform movements and their shape.

SECONDARY OUTCOMES:
ABILHAND-KIDS | 12 weeks
  t evaluates hand skills in children with CP according to the activity frames of ICF-CY. It consists of 21 items. The highest score is 20, the lowest score is 0.
Shriners Hospital Upper Extremity Evaluation (SHUEE) | 12 weeks
  SHUEE is an assessment developed to measure upper extremity function in children with hemiplegic cerebral palsy. SHUEE is a video-based assessment administered by an occupational therapist using standardized objects and tasks. The evaluation takes about 15 minutes.
Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL) | 12 weeks
  This instrument is useful for evaluating interventions designed to improve the lives of children.
Pediatric Evaluation of Disability Inventory (PEDI) | 12 weeks
  Pediatric Evaluation of Disability Inventory assesses key functional capabilities and performance in children ages 6 months to 7 years. PEDI is also useful for older children whose functional abilities are lower than those of seven-year-olds without disabilities.

OTHER OUTCOMES:
Joint Range of Motion (ROM) Measurement | 12 weeks
  Individuals' ROM degrees will be evaluated before and after the treatment using a electronic goniometer in the supine position. Individuals' shoulder flexion, abduction, internal and external rotation, elbow and wrist flexion and extension painless active ROM measurements will be evaluated and recorded.
Modified Tardieu Scale | 12 weeks
  Tardieu is a scale for measuring spasticity that takes into account resistance to passive movement at both slow and fast speed.

CONTACTS AND LOCATIONS:
Overall Officials: AYSE ZENGIN ALPOZGEN, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camden C, Pratte G, Fallon F, Couture M, Berbari J, Tousignant M. Diversity of practices in telerehabilitation for children with disabilities and effective intervention characteristics: results from a systematic review. Disabil Rehabil. 2020 Dec;42(24):3424-3436. doi: 10.1080/09638288.2019.1595750. Epub 2019 Apr 12. PMID 30978110